CLINICAL TRIAL: NCT02598596
Title: Tolerization Reduces Intolerance to Pegloticase and Prolongs the Urate Lowering Effect
Acronym: TRIPLE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ampel BioSolutions, LLC (Industry)
Collaborators: IND 2 Results LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AMP-001
Record Dates: First submitted 2015-10-30; First posted 2015-11-06 (Estimated); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Gout
Keywords: Refractory gout; Chronic gout
MeSH Terms: conditions — Gout | interventions — Pegloticase; Azathioprine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Pegloticase regimen <120 kg - Main Study (Experimental): Subjects weighing <120 kg will receive a tolerizing dose of pegloticase 8 mg IV weekly for the first 3 weeks of dosing followed by an 8 mg IV dose every 2 weeks for a total of 10 doses.
  Interventions: Biological: Pegloticase
- Pegloticase regimen ≥120kg (Experimental): Subjects weighing ≥ 120 kg will be sequentially assigned to 1 of 3 different loading doses (8, 12, and 16 mg) on Study Day 1, and then receive 8 mg on Week 2 and 3, followed by 8 mg every 2 weeks through Week 17 for a total of 10 doses.
  Interventions: Biological: Pegloticase
- Pegloticase PK Sub-Study (Experimental): Subjects weighing <120 kg and ≥120 kg will be assigned to 1 of 2 different loading doses (12 and 16 mg) on Study Day 1, and then receive 8 mg on Week 2 and 3, followed by 8 mg every 2 weeks through Week 17 for a total of 10 doses. Subjects will have multiple blood sampled for PK levels over the 17 week dosing period.
  Interventions: Biological: Pegloticase
- Pegloticase Imaging Sub-Study (Experimental): A subset of subjects participating in the Main Study and weighing <120 kg will have dual-energy computed tomography (DECT) and dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) performed at Screen and at Week 17.
  Interventions: Biological: Pegloticase
- Pegloticase FDG-PET-CT Sub-Study (Experimental): A subset of subjects participating in the Main Study and weighing <120 kg will have fluorodeoxyglucose-positron emission tomography (FDG-PET-CT) to evaluate carotid and aortic (chest) atherosclerosis at Screen and at Week 17.
  Interventions: Biological: Pegloticase
- Pegloticase and Azathioprine (Experimental): Subjects weighing <120 kg will receive azathioprine (AZA) daily for a 2-week run-in period, followed by daily AZA plus pegloticase 8 mg IV every 2 weeks through Week 25 for a total of 13 doses.
  Interventions: Biological: Pegloticase; Drug: Azathioprine

INTERVENTIONS:
Biological: Pegloticase — Pegloticase, IV
  Other Names: Krystexxa
Drug: Azathioprine — Azathioprine (1.25 mg/kg, followed by 2.5 mg/kg) oral, daily
  Other Names: Imuran
  Arms: Pegloticase and Azathioprine

SUMMARY:
The purpose of this study is to evaluate the effect of a high zone tolerizing regimen of pegloticase on clinical outcome, as defined by an serum uric acid level <6 mg/dL, in patients with chronic, refractory gout.

DETAILED DESCRIPTION:
This is an exploratory open-label, multicenter study to evaluate the effectiveness of a 16-week high zone tolerance regimen of pegloticase on response to therapy (serum uric acid <6 mg/dL) with this drug in adult hyperuricemic patients with gout refractory to conventional therapy.

Eligible subjects will receive 1 of 3 different loading doses (8, 12, and 16 mg) on Study Day 1, and then receive 8 mg on Week 2 and 3, followed by 8 mg every 2 weeks through Week 17 for a total of 10 doses.

Subjects will be monitored for efficacy and safety endpoints through Week 17. Subjects will also have blood drawn for pegloticase levels prior to each dose on Weeks 2, 3, 5, 7, 9, 11, 13,15, and 17. Following Study Week 17, subjects will have an option to continue dosing for an additional 8 weeks.

A subset of subjects will participate in additional pharmacokinetic (PK) assessments.

The study duration, per enrolled patient, will be approximately 26 weeks including a 2-week screening period, a 16-week treatment period (end of treatment [EOT] visit Week 17), and an optional 8-week dosing extension.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (age ≥18 years) men and women of non-childbearing potential, with chronic gout refractory to conventional therapy, defined as patients who have failed to normalize SUA and whose signs and symptoms are inadequately controlled with xanthine oxidase inhibitors at the maximum medically appropriate dose, or for whom these drugs are contraindicated.
2. Hyperuricemic - Screening visit SUA must be >6 mg/dL
3. On gout flare prophylactic regimen for 7 days prior to the first dose.
4. Willing and able to give informed consent and adhere to visit/protocol schedules (informed consent must be given before the first study procedure is performed)

Exclusion Criteria:

1. Glucose-6-phosphate dehydrogenase (G6PD) deficiency (confirmed at Screening visit)
2. Non-compensated congestive heart failure, uncontrolled arrhythmia, treatment for acute coronary syndrome (ACS) (myocardial infarction or unstable angina) or hospitalization for congestive heart failure within 3 months of screening or uncontrolled blood pressure (>160/100 mm Hg) at baseline (Screening and pre-dose at Week 1 visit )
3. Women of childbearing potential defined as:

   * Pre- or perimenopausal (<24 months of natural [spontaneous] amenorrhea).
   * <6 weeks after surgical bilateral oophorectomy with or without hysterectomy.
4. Prior treatment with pegloticase or another recombinant uricase
5. Prior treatment or concomitant therapy with a polyethylene glycol (PEG) conjugated drug
6. Known allergy to PEG products or history of anaphylactic reaction to a recombinant protein or porcine product
7. Concurrent treatment with urate lowering agents (ULAs), such as allopurinol and febuxostat. Patients treated with these medications must discontinue treatment 7 days prior to the first dose of study drug
8. Recipient of an investigational drug within 4 weeks prior to study drug administration or plans to take an investigational agent during the study
9. Current liver disease as determined by alanine transaminase (ALT) or aspartate transaminase (AST) levels >3 times upper limit of normal (ULN)
10. History of malignancy within 5 years other than basal cell skin cancer or carcinoma in situ of the cervix
11. Has any other medical or psychological condition which, in the opinion of the Investigator, might create undue risk to the patient or interfere with the patient's ability to comply with the protocol requirements, or to complete the study
12. Solid organ transplant recipients
13. Uncontrolled hyperglycemia with a plasma glucose value >240 mg/dL at screening
14. Currently on dialysis

    Additional Exclusion Criteria for Imaging Sub-study Only
15. Contraindication to receiving a gadolinium-based contrast agent (GBCA) or > 2 previous lifetime exposures to a GBCA
16. Implanted pacemaker, certain older intracranial aneurysm clips, cochlear implants, certain prosthetic devices, implanted drug infusion pumps, neurostimulators, bone-growth stimulators, certain intrauterine contraceptive devices, or any other type of iron-based metal implants.
17. Any internal metallic objects such as bullets or shrapnel, as well as most surgical clips, pins, plates, screws, metal sutures, or wire mesh.

    Additional Exclusion Criteria for FDG-PET-CT Sub-study Only
18. Contraindication to FDG

    Additional Exclusion Criteria for Pegloticase and AZA Therapy Arm Only
19. Any active serious bacterial infection (2 weeks prior to screening) requiring antibiotic treatment
20. Severe chronic or recurrent bacterial infections, such as recurrent pneumonia, chronic bronchiectasis
21. Current immunocompromised condition, including current or chronic treatment with systemic immunosuppressive agents (e.g., prednisone or equivalent dose >510 mg/day)
22. At risk for tuberculosis. Specifically, subjects with: a) current clinical, radiographic, or laboratory evidence of active or latent tuberculosis; b) a history of active tuberculosis within the last 31 years even if it was treated; c) a history of active tuberculosis >31 years ago unless there is documentation that the prior anti-tuberculosis treatment was appropriate in duration and type
23. Known history of hepatitis B surface antigen-positivity or hepatitis B DNA positivity
24. Known history of hepatitis C RNA-positivity
25. Known history of human immunodeficiency virus positivity
26. Severe chronic renal impairment (glomerular filtration rate <25 mL/min/1.73 m2)
27. AZA treatment is contraindicated or considered inappropriate
28. Subject has a homozygous or heterozygous thiopurine methyltransferase (TPMT) variant genotype
29. Diagnosis of osteomyelitis
30. Known hypoxanthine-guanine phosphoribosyl-transferase deficiency, such as Lesch-Nyhan and Kelley-Seegmiller syndrome
31. Concurrent use of a xanthine oxidase inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2020-04-13 (Actual); Study Completion 2020-04-27 (Actual)

PRIMARY OUTCOMES:
Normalization of serum uric acid (SUA) in subjects receiving a tolerizing regimen of pegloticase | Week 17
  Determine response rate; the last 3 consecutive levels of SUA must be <6 mg/dL
Normalization of serum uric acid (SUA) in subjects receiving pegloticase and azathioprine (AZA) immunosuppressive therapy | Week 25
  Determine response rate; the last 3 consecutive levels of SUA must be <6 mg/dL

SECONDARY OUTCOMES:
Change from baseline in SUA to end of Treatment | Baseline and Week 17
  Change from baseline
Change from baseline in SUA to end of Treatment | Baseline and Week 25
  Change from baseline - AZA arm
Proportion of subjects with SUA <5 mg/dL | Week 17
  Proportion of subjects
Proportion of subjects with SUA <5 mg/dL | Week 25
  Proportion of subjects - AZA arm
Proportion of subjects with SUA <2 mg/dL | Week 17
  Proportion of subjects
Proportion of subjects with SUA <2 mg/dL | Week 25
  Proportion of subjects - AZA arm
Infusion reactions (IRs) and anaphylaxis | Week 17
  Incidence - AZA arm
Infusion reactions (IRs) and anaphylaxis | Week 25
  Incidence
Incidence of anti-pegloticase antibodies | Week 17
  Anti-pegloticase antibodies
Incidence of anti-pegloticase antibodies | Week 25
  Anti-pegloticase antibodies - AZA arm
Mean titer of anti-pegloticase antibodies | Week 17
  Anti-pegloticase antibodies
Mean titer of anti-pegloticase antibodies | Week 25
  Anti-pegloticase antibodies AZA arm
Incidence of gout flares, adverse events (AEs), serious AEs (SAEs), and early terminations due to AEs | Week 17
  Incidence
Incidence of gout flares, adverse events (AEs), serious AEs (SAEs), and early terminations due to AEs | Week 25
  Incidence - AZA arm

OTHER OUTCOMES:
Relationship in change from baseline in SUA from baseline with rate of infusion reactions | Baseline to Week 17
  Correlation between change in SUA and infusion reactions
Relationship in change from baseline in SUA from baseline with rate of infusion reactions | Baseline to Week 25
  Correlation between change in SUA and infusion reactions - AZA arm
Compare trough pegloticase levels | Week 17
  Descriptive statistics
Compare trough AZA levels | Week 25
  Descriptive statistics
Ability of imaging to monitor treatment response | Baseline and Week 17
  To compare the ability of dual-energy computed tomography (DECT) and dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) to monitor treatment response, in a subset of subjects weighing < 120 kg
Evaluate change from baseline carotid and aortic (chest) atherosclerosis | Baseline and Week 17
  Change from baseline as measured by fluorodeoxyglucose-positron emission tomography (FDG-PET-CT), in a subset of subjects weighing < 120 kg
Cmax of pegloticase in subjects weighing ≥ 120 kg and < 120 kg | Up to Week 17
  PK parameter
Tmax of pegloticase in subjects weighing ≥ 120 kg and < 120 kg | Up to Week 17
  PK parameter
AUC of pegloticase in subjects weighing ≥ 120 kg and < 120 kg | Up to Week 17
  PK parameter
Terminal phase half-life of pegloticase in subjects weighing ≥ 120 kg and < 120 kg | Up to Week 17
  PK parameter
CL of pegloticase in subjects weighing ≥ 120 kg and < 120 kg | Up to Week 17
  PK parameter
Vss of pegloticase in subjects weighing ≥ 120 kg and < 120 kg | Up to Week 17
  PK parameter
Accumulation Ratio (AR) of pegloticase in subjects weighing ≥ 120 kg and < 120 kg | Up to Week 17
  PK parameter

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - University of Alabama at Birminingham, Birmingham, Alabama
  - Rheumatology Associates of North Alabama, Huntsville, Alabama
  - The Center for Rheumatology and Bone Research, Wheaton, Maryland
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Saint Paul Rheumatology, Eagan, Minnesota
  - Buffalo Rheumatology and Medicine, Orchard Park, New York
  - Montefiore Medical Center, The Bronx, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - ACME Research, LLC, Orangeburg, South Carolina